CLINICAL TRIAL: NCT01786447
Title: Biomarkers of Brain Injury: Magnitude and Outcome of Mild and Moderate TBI
Status: Terminated | Type: Observational
Sponsor: Banyan Biomarkers, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ATO-04a
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Traumatic Brain Injury: Patients who present to the health care facility with mild or moderate traumatic brain injury (Glasgow Coma Scale 9-15) within 4 hours of injury
- Orthopedic Control: Patients who present to the health care facility with isolated extracranial orthopedic injury within 4 hours of injury

SUMMARY:
The purpose of this study is to determine if specific brain injury biomarkers have utility as blood-based traumatic brain injury (TBI) diagnostic and monitoring tools. This will be accomplished by examining the relationships between potential serum-based TBI biomarkers and clinical measures of injury severity, occurrence of complications, and outcome, in subjects with mild or moderate TBI as well as in orthopedic control subjects.

ELIGIBILITY:
Mild/Moderate TBI Group

Inclusion Criteria:

1. 18 years or older
2. GCS 9-15
3. CT scan as part of clinical evaluation
4. experienced some level of altered mental state at time of injury
5. determination of study eligibility within 4 hours of injury

Exclusion Criteria:

1. Pregnant females
2. Prisoners
3. Anemia or significant blood loss (hemoglobin < 12 mg/dL and/or hematocrit < 35%, and/or clinical state requiring resuscitation with more than 6L of colloid or crystalloid fluid)
4. no clear history of trauma as primary event
5. previous history of stroke, or head injury requiring hospitalization
6. dementia or psychotic illness or neurological condition which may affect outcome
7. unable to speak or understand English

Orthopedic Control Group

Inclusion Criteria:

1. 18 years or older
2. Isolated extracranial orthopedic injury, including fractures
3. Stable vital signs on presentation to ED (pulse < 100bpm and systolic blood pressure > 100 mmHg)

Exclusion Criteria:

1. evidence of brain injury, including abnormal neurological examination, alteration in consciousness, memory or mental status, headache, dizziness, or vomiting following injury
2. not enrolled within 4 hours of injury
3. Pregnant females
4. Prisoners
5. Anemia or significant blood loss (hemoglobin < 12 mg/dL and/or hematocrit < 35%, and/or clinical state requiring resuscitation with more than 6L of colloid or crystalloid fluid)
6. previous history of stroke, or head injury requiring hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who present to the health care facility with either Traumatic Brain Injury (GCS 9-15) or isolated extracranial orthopedic injury within 4 hours of injury
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Assessment of biomarkers to identify patients with TBI from orthopedic controls | 4 hours

SECONDARY OUTCOMES:
Assessment of biomarkers to identify patients with brain lesions on CT scan | 4 hours

OTHER OUTCOMES:
Assessment of biomarkers to identify patients with acute post-injury alterations in mental status | 96 hours
Assessment of biomarkers to identify patients that may have longer-term post-injury neurological deficits using neuropsychological assessments | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Jackson Streeter, MD, Study Chair — Banyan Biomarkers
Locations (1):
- Wayne State University, Detroit, Michigan, United States